CLINICAL TRIAL: NCT05872893
Title: Continuous Infusion of First-Generation 5-HT3 Receptor Antagonists in Combination With Dexamethasone. Can This Modality Improve the Antiemetic Effect
Brief Title: Continuous Infusion of First-Generation 5-HT3 Receptor Antagonists in Combination With Dexamethasone
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immune Oncology Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: IMMONC0009
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms | interventions — Ondansetron; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Each patient will serve as his or her own control. Study participants will be randomly assigned to the sequence of treatment. If the patient is assigned to the experimental arm during the first cycle of chemotherapy, he or she will receive the comparator treatment during the second cycle and vice versa. Treatment modalities will follow each other throughout the whole study period.
  Mean nausea score during each chemotherapy cycle will be calculated. To achieve statistically significant results, 140 chemotherapy cycles must be included in the analysis.
Who Masked: Participant
Masking Description: The experimental group will receive intravenous push injections of 0.9% sodium chloride before each infusion, and the control group will receive a 4-hour infusion of sodium chloride after each dose of push injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ondansetron + dexamethasone, continuous infusion (Experimental): Patients will receive a continuous infusion of age-adjusted doses of first-generation 5-HT3 receptor antagonist ondansetron in combination with dexamethasone
  Interventions: Drug: Ondansetron; Drug: Dexamethasone
- ondansetron + dexamethasone, push injection (Active Comparator): Patients will receive standard i/v push injections of first-generation 5-HT3 receptor antagonist ondansetron and dexamethasone
  Interventions: Drug: Ondansetron; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ondansetron — Patients will receive age-adjusted doses of ondansetron 5mg/m2
Drug: Dexamethasone — Patients will receive dexamethasone 4mg/m2

SUMMARY:
Chemotherapy-induced nausea and vomiting are serious side effects of cancer treatment that can have a significant negative impact on a patient's quality of life. Although the prevalence of nausea and vomiting has significantly decreased due to the implementation of new antiemetic drugs, several studies revealed that approximately 30% to 60% of patients still complain of acute or delayed chemotherapy-induced emesis. It is estimated that slow infusion of ondansetron in combination with dexamethasone can provide long-lasting stable concentrations of drugs in the blood serum contributing to better effect development. Therefore, the investigators suggest a continuous infusion of the above-mentioned drug combination as an alternative with potential superior activity.

DETAILED DESCRIPTION:
Chemotherapy-induced nausea and vomiting are serious side effects of cancer treatment that can have a significant negative impact on a patient's quality of life. It is estimated that 70-80% of patients receiving different chemotherapy regimens can experience emesis. Although the prevalence of nausea and vomiting has significantly decreased due to the implementation of new antiemetic drugs, several studies revealed that approximately 30% to 60% of patients still complain of acute or delayed chemotherapy-induced emesis. Currently, the three categories of drugs with the highest therapeutic index for preventing chemotherapy-induced nausea and vomiting are 5-HT3 receptor antagonists, NK1 receptor antagonists, and glucocorticoids (particularly Dexamethasone). Second-generation 5-HT3 receptor antagonists and NK1 receptor antagonists are more effective due to their prolonged influence but are very expensive and not available in the majority of resource-limited settings. Moreover, NK1 receptor antagonists are not still widely recommended for use in children < 12 years of age. First-generation 5-HT3 receptor antagonists in combination with Dexamethasone have proven superior activity compared to single agents. It is estimated that slow infusion of the above-mentioned agents can provide long-lasting stable concentrations of drugs in the blood serum contributing to better effect development. It has been shown that Ondansetron continuous infusion has superior efficacy in preventing postsurgical nausea and vomiting. Therefore, the investigators suggest a continuous infusion of first-generation 5-HT3 receptor antagonists in combination with Dexamethasone as an alternative with potential superior activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 1 day to 18 years who are diagnosed with cancer and are eligible for chemotherapy.
* Voluntarily agree to participate by giving written parental permission and child assent.
* Patients with sufficient cardiac function, as determined by the investigator.

Exclusion Criteria:

* Patients with a history of severe hypersensitivity reactions or anaphylaxis related to the use of 5-HT3 receptor antagonists.
* Patients receiving concurrent chemo-radiation therapy.
* Patients diagnosed with cardiac arrhythmias and congenital long QT interval syndrome.
* Known clinically significant drug interactions between chemotherapeutic agents and 5-HT3 receptor antagonists and/or Dexamethasone (e.g. more than 0.8 mg/ml concentrations of 5-fluorouracil may cause precipitation of ondansetron).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Mean nausea score per patient | 20 months
  Mean nausea score will be calculated as a weighted average of the Visual Analogue Scale (VAS) or Baxter Animated Retching Faces (BARF) scale observations during each cycle of chemotherapy.

SECONDARY OUTCOMES:
Correlation between mean nausea score and demographic variables | 20 months
Correlation between mean nausea score and disease characteristics | 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Julieta Hoveyan, MD, Principal Investigator — Immune Oncology Research Institute; Ruzanna Papyan, MD, Study Chair — Immune Oncology Research Institute; Samvel Bardakhchyan, MD, PhD, Study Chair — Immune Oncology Research Institute; Gevorg Tamamyan, MD, PhD, DSc, Study Director — Immune Oncology Research Institute
Locations (1):
- Hematology Center named after prof. R. Yeolyan, Yerevan, Armenia